CLINICAL TRIAL: NCT05549778
Title: Safety and Efficacy of the Stomach Ulcer Drug Polaprezinc (POL) on Enzalutamide- or Abiraterone-resistant CRPC
Brief Title: Polaprezinc Treatment for Enzalutamide- or Abiraterone-resistant CRPC
Acronym: PEACe
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangnan University (Other)
Collaborators: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JiangnanU RWang-2
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-05

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: CRPC; POL
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients will be on abiraterone/prednisone plus polaprezinc, or with other treatments according to patients'wishes in consultation with physicians.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polaprezinc group (Experimental): Patients will be on abiraterone plus polaprezinc (75 mg b.i.d. for 6 months)
  Interventions: Drug: Polaprezinc group
- Control group (Active Comparator): Patients will be on abiraterone, radiotherapy or chemotherapy for 6 months
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Polaprezinc group — Abiraterone plus Polaprezinc for 6 months
  Other Names: POL
  Arms: Polaprezinc group
Drug: Control group — Abiraterone, radio- or chemotherapy
  Other Names: OTH
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate clinical safety and efficacy of a gastric ulcer drug, polaprezinc (POL), with the AR-inhibitor abiraterone in Chinese patients with castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
Prostate cancer (PCa) is a major disease that affects 14.1% male population worldwide with a 6.8% mortality rate in 2020 (https://gco.iarc.fr/). In China, the PCa incidence rate is lower than in Europe and the US but increases rapidly. Androgen deprivation therapy (ADT) has been the most used treatment for men with advanced prostate cancer for decades. Despite the initial favorable response, nearly all patients progress to castration-resistant prostate cancer (CRPC) and subsequently succumb to the disease within 1-3 years.

Zinc-L-carnosine (ZnC), also called polaprezinc (otherwise known as PepZin GI™), is a chelated compound that contains L-carnosine and zinc. Some reports indicated that POL is effective in restoring the gastric lining, healing other parts of the gastrointestinal (GI) tract, improving taste disorders, improving GI disorders, and enhancing skin and liver. The primary mechanisms of POL action are identified as anti-inflammatory and antioxidant pathways. We have identified PRDX5 as a therapeutic target and repurposed polaprezinc (POL) as its inhibitor for the treatment of CRPC.

CRPC patients will be enrolled with their fully informed consent. Patients will be on abiraterone/prednisone, abiraterone/prednisone plus polaprezinc granules, or with other treatments according to patients' wishes in consultation with physicians. Polaprezinc will be 75 mg b.i.d., for 6 months. A standard regimen will be used for other treatments. PSA will be measured every month. ECT will be taken before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients were older than 18 years of age.
2. Patients with measurable disease were required to have documented disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) (28) with at least one bone metastatic lesion. Patients with non-measurable disease were required to have at least two consecutive increases (relative to a reference value measured at least a week apart) in serum PSA.
3. Patients had been taking abiraterone or enzalutamide for at least three consecutive months and showed a persistent rise in PSA.
4. Life expectancy >6 months

Exclusion Criteria:

1. Patients had taken polaprezinc previously.
2. Patients had cancer therapy (other than ADT) within 4 weeks before enrolment.
3. Patients had malignancies other than prostate cancer.
4. Patients had uncontrolled severe illness or medical conditions.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
PSA response | 6 months
  Decrease in PSA level or slowdown in PSA progression
Disease progression | 6 months
  Non-progressive disease (Non-PD) by ECT imaging analysis according to the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yong Q Chen, MD/PHD, Principal Investigator — Jiangnan University
Locations (1):
- Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No